CLINICAL TRIAL: NCT02876276
Title: Minimally Invasive Treatment for Papillae Deficiencies in Esthetic Zone Using Hyaluronic Acid
Brief Title: Hyaluronic Acid in Papillary Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_36683
Record Dates: First submitted 2016-08-12; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Interdental Papillary Reconstruction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- HA filler group (Active Comparator): 6 weeks after the initial therapy, patients were scheduled for the procedure.16 Local Anesthetic solution (2% Lignocaine HCl with adrenaline 1:80000) was administered.17 About 0.2 ml of a commercially available hyaluronic acid based gel was injected 2-3 mm coronal to the apical tip of the receded interdental papilla . Injections were performed using 23 gauge X 25mm intraoral injection needles . The concentration of HA gel used was 20 mg/ml.6 The area was gently massaged to ensure that the filler was uniformly distributed. Care was taken to fill each papilla to full correction (100% of defect). After the treatment the individual patient syringes were capped and stored in a refrigerator with patient names and details. The needle was discarded. Patients were seen three weeks after the initial treatment and if augmentation was still deemed necessary, another injection of 0.2ml was injected up to three times
  Interventions: Procedure: Hyaluronic acid filler
- saline filler group (Placebo Comparator): with saline same protocol was performed as mentioned in test group
  Interventions: Procedure: Hyaluronic acid filler

INTERVENTIONS:
Procedure: Hyaluronic acid filler — Papillary augmentation with HA dermal fillers was considered as the test group

SUMMARY:
Hyaluronic acid (HA) has been used as a dermal filler in medicine for many years. It also has umpteen benefits in terms of aiding in rapid healing and resolution of inflammation. Thus in the present study, HA has been used at the test site to fill papillary recession defects. At the control site saline was injected as the placebo.

DETAILED DESCRIPTION:
INTRODUCTION Periodontal diseases, trauma, treatment of periodontal diseases and iatrogenic causes lead to papillary tissue loss in the interproximal area.1 Management of soft tissue deformities in the interproximal space can be advocated through several surgical and non-surgical techniques. The non-surgical approaches - orthodontic, prosthetic and restorative procedures modify the interproximal space, thereby altering the soft tissue morphology. The surgical techniques aim to recontour, preserve or reconstruct the soft tissue between teeth and implants. Surgical techniques, due to their invasive and unpredictable nature and limited blood supply/ minimal access makes regeneration of deficient papilla a highly sensitive procedure.2 Hyaluronic acid (HA) is a high molecular weight polysaccharide that plays a vital role in the functioning of extracellular matrices, including those of mineralized and non-mineralized periodontal tissues. HA helps in tissue hydrodynamics, cell migration/ proliferation, anti-inflammatory role and facilitates healing.3 HA has shown anti-inflammatory, anti-edematous and anti-bacterial effects in the treatment of gingivitis and periodontitis.4 Deviating from these utilities, HA also plays an important role in the non surgical facial rejuvenation through bioengineered hyaluronic acid derivatives. The exquisite role of bioengineered hyaluronic acid derivatives for soft tissue augmentation in gingival deficiencies has not been researched enough. Based on this beneficial effect of HA in dermatology, the present triple blind split mouth randomised clinical trial was planned to evaluate the injection of HA dermal filler as a minimally invasive treatment modality for the reconstruction of lost interdental papilla.

The aim of the present study was to evaluate the efficacy of hyaluronic acid dermal filler for interproximal papillary augmentation in Nordland's Class I and Class II5 interdental papillary recession defects.

MATERIALS AND METHODS:

PARTICIPANTS:

15 adult patients from the out-patient department of Department of Periodontology, Krishnadevaraya College of Dental Sciences, Bangalore, India, aged between 25-75 years were recruited among those seeking treatment for esthetics in the maxillary anterior region due to interdental papilla recession, from July 2013 to September 2014. The details of the study and the procedure were explained to the patients and an institutional review board approved informed consent was obtained from each patient, affiliated to Rajiv Gandhi University of Health Sciences (ACA/DCD/SYN/KCODS - B/PG/2012-2013) (02_D012_36683).

INTERVENTIONS Papillary augmentation with HA dermal fillers was considered as the test group and this was compared with saline injection (placebo) for the control group. The study was conducted in full accordance with the declared ethical principles (World Medical Association Declaration of Helsinki, version VI, 2002) and was approved by the Institutional review board of Krishnadevaraya College of Dental Science and Hospital, affiliated to Rajiv Gandhi University of Health Sciences, Bangalore.

This study was conducted by 2 investigators and one operator, one of the investigators and the operator were blinded. The unblinded investigator performed the randomisation and allocation of the test and control groups, whereas all the study measurements and assessment were performed by the blinded investigator and operator. The patients were not informed and had no way to decipher the test or the control group. Both the investigators assessed the following clinical outcomes.

STUDY DESIGN The design of this study is a unicenter, triple blind, placebo controlled split mouth randomised controlled clinical trial according to the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010 (Fig 1). All patients completed an initial therapy that included oral hygiene instructions and scaling and root planning. 2 similar sites in each patient i.e. a total of 30 interdental papillary recession area were selected and treated. One of the patients failed to complete the follow up visits and hence was excluded from the study.

DATA COLLECTION Data collection included baseline clinical measurements and photographs taken perpendicular to the site at baseline, 3 weeks, 3 months and 6 months.

The radiographs were taken using a positioning device and an intraoral periapical radiograph grid at baseline and 6 months. Study impressions of sites were taken at baseline.2 At baseline and all subsequent study visits the below mentioned clinical parameters were recorded by the examiner using a standardized acrylic stent and University of North Carolina (UNC 15) probe , i.e. papillary recession depth (distance from the contact point to gingival margin was measured to the nearest millimeter- CP -GM); Interproximal width (distance from the mesial height of contour to the distal height of contour of the interproximal tissue-IPW); Width of the keratinized gingiva (schiller's potassium iodide solution-KTW); Facial gingival recession of the two adjacent teeth11; Radiographic Analysis of papillae height (vertical distance from the tip of the interdental papillae, using radiopaque material to mark it to the tip of the crest of the alveolar bone)12; Plaque index (PI)13; Gingival Bleeding Index (GBI)14; Gingival Index (GI)15 and photographic analysis of the intraoral photographs taken using Image analysis software. (Digimiser∗)6

OUTCOMES:

Two different treatment methods were compared, HA filler (n=15) and saline (n=15). The primary outcome that was assessed in the study was the papillary recession reduction (pRecRed). pRecRed was calculated in millimeters and in percentage papillary coverage(PPC). The percentage of complete papillary coverage (CPC) in each group was assessed.

The formula used to calculate the percentage papillary coverage was as follows-

Baseline (CP-GM) - 6 month (CP-GM)

---------------------------------------------- x 100 Baseline (CP-GM) The primary outcomes were also assessed with a photogrammetric analysis using Digimiser software∗. Image analysis consisted of several steps: image identification, image scaling, calibration, and measurement. The ideal image was selected and scaled to standard (1:1) magnification. The photograph was calibrated and standardised to the actual clinical dimensions by feeding a known clinical dimension (the 1mm markings of UNC-15∗∗∗periodontal probe in the photograph) into the software. Determination of the distance from the contact point to the gingival margin was done (CP-GM) .The ideal height of the interdental papillary recession was measured as the distance between the lines joining the apical tip of the papilla to the contact point of the teeth. The primary outcome measurement i.e. papillary recession depth was assessed using the computerized software tools.

The following secondary outcomes were also measured change in interproximal width2; width of the keratinized gingiva9; facial gingival recession of the two adjacent teeth11; radiographic height of papillae height using12; Plaque index13; Gingival Bleeding Index14 and Gingival Index15.

PRE-TREATMENT PROCEDURES:

Initial therapy that included scaling and root planning was completed prior to the treatment procedure.10 The patients who demonstrated ≤ 20 % O'Leary Plaque Index were subjected to the study protocol.2 Occlusal interferences were identified and eliminated through occlusal adjustments, and hard acrylic bite guards were constructed for those patients with parafunctional habits. The study was designed so that extraneous factors such as oral hygiene and compliance were controlled within each subject.

RANDOMIZATION:

Randomization sequence was generated by a computer program. Allocation concealment was achieved using a sealed coded opaque envelope containing the treatment of the specific subject. The unblinded investigator opened the sealed envelope containing treatment assignment as Test site (treatment with HA filler) or Control Site (treatment with placebo) prior to the treatment procedure and allotted the cases to operator accordingly. The patient and investigator and operator were blinded to the treatment performed.

PROCEDURE:

6 weeks after the initial therapy, patients were scheduled for the procedure.16 Local Anesthetic solution (2% Lignocaine HCl with adrenaline 1:80000) was administered.17 About 0.2 ml of a commercially available hyaluronic acid based gel was injected 2-3 mm coronal to the apical tip of the receded interdental papilla (Fig 2). Injections were performed using 23 gauge X 25mm intraoral injection needles . The concentration of HA gel used was 20 mg/ml.6 The area was gently massaged to ensure that the filler was uniformly distributed. Care was taken to fill each papilla to full correction (100% of defect). After the treatment the individual patient syringes were capped and stored in a refrigerator with patient names and details. The needle was discarded. Patients were seen three weeks after the initial treatment and if augmentation was still deemed necessary, another injection of 0.2ml was injected up to three times.6 In the control site the same protocol was performed, however with saline. Patients were recalled and all the clinical and radiographic parameters were recorded after three months and six months.

SATATISTICAL ANALYSIS:

A sample of 14 recessions in each group (test and control), were included. The analysis was performed by a blind examiner. Statistical analysis was undertaken with SPSS (version10.0.5) package. Normality of data was tested using Shapiro-Wilk test. The intergroup comparisons were done using student 't' test and chi square test, with Mann Whitney U test as post hoc test. Intergroup comparison at different recall visits was done using Mann Whitney U test. The intergroup comparison of the photogrammetric analysis; mean papillary recession reduction between test and control at baseline and 6 months was compared using student 't' test with Mann Whitney U test as post hoc test. Intragroup comparison between baseline and the follow up visits values were done using the one was ANOVA test and Kruskal Wallis test. Comparison between the clinical analysis and image analysis was done using chi square test.

DISCUSSION The attempt to use dermal fillers for papillary augmentation is scarcely reported in the existing literature. Only one study has evaluated the effect of HA filler on interdental papilla reconstruction and noted that injection of hyaluronic acid gel is safe and significantly decreased the interdental black triangle in the esthetic zone.3 Application of non-invasive techniques such as the use of commercially available hyaluronic acid gel can replace the conventional invasive methods.

This split mouth clinical study consisted of 15 patients with Nordland and Tarnow's Class I and Class II6 papillary loss that were treated with either HA gel (test) or saline (control) for papillary augmentation.

Significantly 28.6% of the sites in test group showed CPC whereas no sites in the control group showed CPC. The results are in agreement with that of Becker et al. 2010 who achieved 21.4% CPC similarly by injection of a HA gel for papillary augmentation.3 CPC was noted by Nordland et al 200818, where he used a microsurgical technique to reconstruct the lost interdental papilla, Tinti C et al. 200219 used Ramp mattress suture to augment the papilla, Carnio et al. 200420 - interposed subepithelial connective tissue graft and Geurs et al10 showed 57.9% of CPC. Various other authors have also reported CPC with different techniques.21-24 55.4% of PPC was achieved with HA augmentation, which is similar to 42.1% PPC achieved by Geurs et al. 201210 who used micronized acellular dermal matrix allograft for papillary reconstruction. Another similar study has shown a significant papillary fill post operatively.2 No significant differences were noted in both the groups as regards to the interproximal width. A similar trend was noted by Mcguire & Scheyer 2007.2 There were no significant changes in the dimensions of the keratinized gingiva in both the groups.

Image analysis system to measure changes in root coverage has also been successfully employed in previous literature.26 Identification of the anatomic CEJ, accuracy of determining the probing pocket depth/ papillary height/ width etc. can be subjected to manual errors. Calibrated photogrammetric analysis can reduce subjective measurement errors. The current study reported no significant differences between clinical and photogrammetric analysis. 26 Literature review reveals that the split mouth randomised controlled clinical trial with a duration of more than or equal to 6 months assessing complete papillary coverage as the primary outcome in papillary reconstruction for papillary recession defects is rarely documented. However, there is frequent reporting of primary outcome variable like PPC, pRecRed, change in papillary index scores and the casual mention of significant papillary gain. Due to the inconsistent and insufficient data available regarding papillary reconstruction, it was difficult to compare the results of the current trial.

Hyaluronic acid gel§§§ is generated by Streptococcus species of bacteria and is chemically cross-linked and has a concentration of 20 mg/mL. Hyaluronic acid fillers are less allergy prone and produce favourable results.27 Hyaluronic acid forms the natural physiological constituent of the ground substance of connective tissue of the gingival mucosa, and hence can be considered for the treatment of papillary deficiency. Patients on blood thinning agents might experience mild bruising, therefore eliminating any blood thinning agents for at least 7 days before injection is preferred.28 HA acts as a matrix, provides lubrication and increases volume through its aqueous and pliable framework that suspends and adheres to collagen, elastin and numerous proteins like fibrinogen, fibrin, fibronectin and collagen bind to HA.29 HA integrates well into the adjacent gingiva with excellent esthetic results. Microcirculatory perfusion is enhanced with HA.30 The plumping of the interdental papilla on injecting the defect with a HA filler could be explained by the fact that HA has a unique rheological property and is highly hydrophilic and can bind to upto 1000 times more water than its molecular-weight.31 HA injection has shown to increase denovo collagen synthesis, hypothesized to be the result of fibroblast stretching. As HA is degraded novel collagen synthesis replaces the HA resulting in longer lasting correction.32 CPC achieved and maintained in the current trial can be attributed to the hydrophilpic nature and collagen synthesizing property of HA filler. The cross linking prevents its degradation in the body. The high level of cross linking alters the ability of water to bind to HA and thereby creates tissue lift.28 HA increases the cell division and the tubulin concentration which helps in the proliferation of fibroblasts through the cell cycle.33 HA also acts as biomaterial scaffold for other molecules, such as BMP-2 and PDGF-BB.4 Smooth-gel dermal fillers like HA offer longer-lasting correction of defects than bovine collagen etc. The insoluble gel portion that persists in the skin and gingiva after injection is the amount of HA that contributes to the clinical effect.34 The product in trial being a smooth gel HA dermal filler offers long lasting correction and achieves natural look post injection.35 Nearly all the subjects achieved optimal correction with only a single injection of 0.2ml of HA dermal filler.6 The commonly employed injection techniques for dermal fillers (serial puncture, linear threading, fanning and cross hatching) was not employed in the current trial owing to the limited area and minimal access to the interdental papillary region. The product that is used in the current study is 1.8% sodium salt hyaluronic acid. It has been successfully used in the treatment of nasolabial folds with no adverse events.36 Results from this study evaluating the use of a commercially available injectable gel for correcting deficient papillae between teeth are successful and promising and minimally invasive. This study had a follow up period of 6 months as compared to the study of Becker et al. 20106 which had a follow up period of 6-25 months based on the patient compliance. It is interesting to note that all patients considered treatment to be painless.

Traditional gingival augmentation uses epithelial/ connective tissue graft harvested from the palate that can cause considerable discomfort for the patient which is successfully avoided with HA dermal filler.

Randomized clinical trials with a longer follow up time period and a larger sample size are to be undertaken to further justify the use of HA dermal filler for the augmentation of papillary deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 25-75 years, with at least one pair of similar bilateral, Nordland's class I and class II loss of interdental papillae in the maxillary anterior region, radiographic evidence of sufficient interdental alveolar bone (i.e. distance between alveolar crest and contact point ≤ 5mm), pocket probing depth ≤ 4mm, systemically healthy patients, patients willing to participate in the study and patients with esthetic concerns

Exclusion Criteria:

* Patients with known allergy to hyaluronic acid, patients with poor plaque control.(≥20% O'Leary plaque index), medically compromised patients, pregnant and lactating women, history of smoking, who had received a crown or pontic on one or both teeth involved in the interproximal space, interproximal spaces next to teeth that included root grooves, furcations, Miller's tooth mobility index >18, open contacts, probing depths >3 mm, and radiographic evidence of pathology, with translocated or tilted teeth, and who had undergone papillary regeneration procedures in the area selected previously

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
the papillary recession reduction (pRecRed). | 6 month
  . papillary recession depth (distance from the contact point to gingival margin was measured to the nearest millimeter- CP -GM)
percentage papillary coverage(PPC | 6 month
  The formula used to calculate the percentage papillary coverage was as follows-
  Baseline (CP-GM) - 6 month (CP-GM)
  ---------------------------------------------- x 100 Baseline (CP-GM)